CLINICAL TRIAL: NCT06027749
Title: Impact of Capturing Ictal Events With Ultra-long-term Ambulatory EEG Monitoring With REMI.
Brief Title: Impact of Capturing Ictal Events With Ultra-long-term Ambulatory EEG Monitoring With Remote EEG Monitoring System.
Acronym: REMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epitel, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REMI-23-01
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy; Seizures
Keywords: EEG Monitoring
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Epitel's™ Remote EEG Monitoring System's (REMI™) — Ambulatory electroencephalography (EEG) monitoring

SUMMARY:
The goal of this clinical trial is to test Epitel's™ Remote EEG Monitoring System's (REMI™) ability to record electroencephalography (EEG) of seizure events in an ambulatory setting for extended periods (14 - 28 days) in patients presenting with questionable seizure characterization. The main questions it aims to answer are: • Can more seizure events be recorded in fourteen (14) days than can be recorded in three (3) days? • Do treating clinicians find clinical value in extended fourteen (14) - twenty-eight (28) days of EEG? Participants will wear a portable EEG device (REMI) for fourteen (14) to twenty-eight (28) days in their home/community setting.

DETAILED DESCRIPTION:
This is a prospective study to quantify Epitel's™ Remote EEG Monitoring System's (REMI™) ability to record electroencephalography (EEG) of seizure events in an ambulatory setting for extended periods (14 - 28 days). Patients presenting with questionable seizure characterization that are scheduling a conventional at home ambulatory EEG (Amb EEG) and who meet the study inclusion and exclusion criteria will be prescribed a REMI system.

The purpose of this study is to demonstrate that the REMI system is able to record EEG data that clinicians can use to identify ictal events over extended periods, and that extended clinical EEG data is valuable in the diagnosis and treatment of seizure related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a reported history of seizures (epileptic, non-epileptic, or unknown),
* Have a minimum reported seizure rate of one every two weeks,
* Are prescribed an ambulatory EEG study as part of routine care,
* Is Male or Female between the ages of 18 and 70,
* Can understand and sign written informed consent, or have a legal guardian provide consent,
* The Patient (or Primary Caregiver) must be competent to follow all study procedures,
* The Patient must be willing to use the System for a prolonged period (up to 30 days), for a minimum of 20 hours/day.

Exclusion Criteria:

* Is sensitive or allergic to medical acrylics, silicones, or hydrogels,
* Is enrolled in another investigational drug or device trial,
* Is homeless or in a home without a power supply, or
* Cannot read, speak, or understand English (and does not have a translator).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Ictal Events Identified in fourteen (14) days. | Fourteen (14) days
  Epileptiform seizure activity as identified by three independent board-certified epileptologists assessing data collected by REMI. The number of seizures identified in the first three days will be compared to the number of seizures identified during days one (1) to fourteen (14).

SECONDARY OUTCOMES:
Extended Use | Twenty-eight (28) days
  Epileptiform seizure activity as identified by three independent board-certified epileptologists assessing data collected by REMI. The number of seizures identified in the first fourteen (14) days will be compared to the number of seizures identified during all twenty-eight (28) days.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.